CLINICAL TRIAL: NCT06087874
Title: Preventive Effect of Perinatal Oral Probiotic Supplementation (POPS) on Neonatal Jaundice: A Randomized Double-Blind Placebo-Controlled Parallel-Group Superiority Clinical Trial
Brief Title: Preventive Effect of Perinatal Oral Probiotic Supplementation (POPS) on Neonatal Jaundice
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ronald Wang, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20230317
Record Dates: First submitted 2023-10-05; First posted 2023-10-18 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Neonatal Jaundice; Microtia; Pregnancy Related; Hyperbilirubinemia, Neonatal
MeSH Terms: conditions — Jaundice, Neonatal; Congenital Microtia; Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: It is a double-blind study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Vivomixx® is a multi-strain probiotics product.
  Interventions: Dietary Supplement: Vivomixx®
- Placebo (Placebo Comparator): Maltose-containing placebo product
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vivomixx® — The probiotic group participants will receive 1 sachet of probiotic product daily from 36weeks of gestation up to 7th day of postpartum while placebo groups will 1 sachet placebo prepared with the same colour, taste, and packaging with Vivomixx® daily for the same duration of probiotic groups. Vivomixx® is a non-genetically modified (GMO), gluten-free, high potency microbiotic food supplement, containing eight strains (Streptococcus thermophilus DSM24731® / NCIMB 30438, Bifidobacterium breve DSM24732® / NCIMB 30441, Bifidobacterium longum DSM24736® / NCIMB 30435, Bifidobacterium infantis DSM24737® / NCIMB 30436*, Lactobacillus acidophilus DSM24735® / NCIMB 30442, Lactobacillus plantarum DSM24730® / NCIMB 30437, Lactobacillus paracasei DSM24733® / NCIMB 30439, Lactobacillus delbrueckii subsp. bulgaricus DSM24734® / NCIMB 30440) of live bacteria (450 billion bacteria per sachet).
  Arms: Probiotics
Dietary Supplement: Placebo — A maltose- containing product with a similar phenotype with Vivomixx®.
  Arms: Placebo

SUMMARY:
This is a randomized double-blind placebo-controlled parallel group superiority clinical trial among 94 pregnant women (47 in each group) to investigate the effect of maternal perinatal probiotic supplementation on neonatal jaundice, breast milk microbiome, maternal stool, and infant fecal microbiome. Vivomixx®-probiotic product will be used as treatment and placebo as a control.

DETAILED DESCRIPTION:
Neonatal jaundice is a yellowish discoloration of the skin and sclera because of over-concentration of circulating unconjugated bilirubin (hyperbilirubinemia) in the body. It can lead the baby to severe complications including death. Intestinal flora modulation by probiotics administration to the mother may tackle this problem. Therefore, investigators designed a randomized double-blind placebo-controlled parallel group superiority clinical trial among 94 pregnant women (47 in each group). Eligible pregnant women will be recruited voluntarily at 28-36 weeks of gestation and allocated randomly to either the probiotic group (Vivomixx®) or placebo group (maltose-containing unit) which are phenotypically similar. Participants will take one sachet of the product per day starting from 36 weeks of gestation until the end of first week of postpartum. Biological samples (maternal stool, breast milk, and neonatal faeces) will be collected at different time points. Additionally, neonatal transcutaneous bilirubin will be measured on the second and seventh day of life using a Drager Meter (a transcutaneous bilirubinometer). The microbial DNA will be extracted from biological samples using commercial kits and metagenomics sequencing will be employed and will be correlated with bilirubin level using appropriate statistical methods. This study will be conducted based on the Helsinki Declaration and International Council for Harmonization Requirements for Pharmaceuticals for Human Use (ICH) Guideline for Good Clinical Practice (GCP) standards. Ethical approval is obtained from the Joint Chinese University of Hong Kong and New Territories East Cluster (CUHK-NTEC) Clinical Research Ethics Committee, Hong Kong with reference number: 2023.100-T. Written informed consent will be obtained from each participant during enrolment.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women aged 18-45 years old.
* Gestational age of 28-34 weeks
* Normal singleton pregnancy

Exclusion Criteria:

* Foetal abnormality
* Mothers with antibiotic medication during the allocation
* Couples with glucose 6-phosphate dehydrogenase enzyme deficiency
* Couples with known rhesus or haemolytic disease history
* Plan of place of birth at other hospitals other than Prince of Wales Hospital
* known breast disorder or any contraindication for breastfeeding.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-03-23 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Hyperbilirubinemia | 1 week since birth
  Investigators will measure the transcutaneous bilirubin level on the second and seventh day of life and plot the record on the nomograph. The record above the 95th percentile will be taken as considerable hyperbilirubinemia and then the baby will be investigated for total serum bilirubin measurement if needed to declare hyperbilirubinemia. The outcome will be classified as hyperbilirubinemia and non-hyperbilirubinemia.
Transcutaneous bilirubin level | 1 week of life (after birth)
  Infant's skin bilirubin level on the chest measured using a non-invasive devise called Drager meter. It will be measured in milligram per decilitre or micromole per liter. This outcome will be measured as a continuous outcome.

SECONDARY OUTCOMES:
Preterm birth | within two days of birth
  This will be measured using the gestational age at birth
Number of participants with Initiation of labor | within two days of birth
  Spontaneous initiation of induction of labour
Mode of birth checklist | within two days of birth
  Spontaneous vaginal delivery, assisted birth or cesarean section
Birth weight | within two days of birth
  Weight of the baby at birth in grams
Apgar scores | within two days of birth
  First and fifth-minute Apgar scores of babies
Breast milk microbiome profile | From birth seventh day of postpartum
  Breast milk samples will be collected, bacterial DNA collected and meta-genomic sequencing will be carried out.
Stool microbiome profile | From birth seventh day of postpartum
  maternal and infant stool samples will be collected, bacterial DNA collected and meta-genomic sequencing will be carried out.

OTHER OUTCOMES:
Number of participants with Skin rash | From initiation of the intervention until 1 week postpartum
  any allergic reaction
Number of participants with Diarrhea | From initiation of the intervention until 1 week postpartum
  Frequent loose of stool
Number of participants with Abdominal bloating | From initiation of the intervention until 1 week postpartum
  Any distention, gas (flatulence) and cramp on the abdomen

CONTACTS AND LOCATIONS:
Overall Officials: Chi C Wang, Professor, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be included in publications of findings as a supplementary file. It will be available to anyone based on official request from the principal investigator.
Supporting Information: Study Protocol
Time Frame: One year after initiation of the study
Access Criteria: official request and memorandum of understanding signing

REFERENCES:
- [Derived] Alemu BK, Lee MW, Leung MBW, Lee WF, Wang Y, Wang CC, Lau SL. Preventive effect of prenatal maternal oral probiotic supplementation on neonatal jaundice (POPS Study): A protocol for the randomised double-blind placebo-controlled clinical trial. BMJ Open. 2024 Jun 8;14(6):e083641. doi: 10.1136/bmjopen-2023-083641. PMID 38851232